CLINICAL TRIAL: NCT00043368
Title: A Continuation Study Of PF-3512676 (CPG 7909) Injection In Patients With Metastatic Or Recurrent Malignancies Who Have Stable Disease Or Who Have Responded To Pf-3512676 Injection Therapy
Brief Title: PF-3512676 (CPG 7909) Injection For Patients Who Completed An Oncology Study Using PF-3512676 (CPG 7909)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C016; CO16, A8501015
Record Dates: First submitted 2002-08-08; First posted 2002-08-12 (Estimated); Last update posted 2009-03-12 (Estimated); Status verified 2009-03

CONDITIONS: Melanoma; Breast Neoplasms; Carcinoma, Renal Cell; Lymphoma, T-Cell; Carcinoma, Non-Small-Cell Lung
Keywords: CPG 7909 continuation study
MeSH Terms: conditions — Melanoma; Breast Neoplasms; Carcinoma, Renal Cell; Lymphoma, T-Cell; Carcinoma, Non-Small-Cell Lung | interventions — ProMune

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Patients will be treated with the same dosing regimen and schedule of PF-3512676 Injection with which they were treated at the end of the previous PF-3512676 Injection trial. Any proposed changes to their schedule/regimen will be at the discretion of the treating physician, following consultation with Coley.
  Interventions: Drug: PF-3512676

INTERVENTIONS:
Drug: PF-3512676 — PF-3512676 IV at doses: 0.01mg/kg, 0.16mg/kg and 0.32mg/kg PF-3512676 Injection given by subcutaneous injection at doses: 0.04mg/kg, 0.16mg/kg, 0.20mg/kg, 0.28mg/kg, 0.32mg/kg, 6mg, 10mg, 40mg.
  Other Names: CPG 7909, ProMune

SUMMARY:
This protocol allows patients who completed Coley oncology studies using PF-3512676 (CPG 7909) Injection to continue receiving the treatment until disease progression.

ELIGIBILITY:
Inclusion Criteria:

Immediate (within 4 weeks) prior completion of a clinical trial of PF-3512676 Injection alone or in combination with other anti-neoplastic treatment for malignancy.

Exclusion Criteria:

The patient has received any anti-neoplastic therapy since completing a prior trial with PF-3512676 Injection, or has participated in another clinical trial following participation in a trial with PF-3512676 Injection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2002-09; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Adverse Events and DLTs will be evaluated by the Investigator and summarized. | indeterminate

SECONDARY OUTCOMES:
No formal statistical analysis of this study will be conducted. All clinical data may be summarized and included in data listings. | indeterminate

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (27):
- United States (26):
  - Pfizer Investigational Site, Berkely, California
  - Pfizer Investigational Site, Gilroy, California
  - Pfizer Investigational Site, Hollister, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Palm Springs, California
  - Pfizer Investigational Site, Stanford, California
  - Pfizer Investigational Site, New Haven, Connecticut
  - Pfizer Investigational Site, Bonita Springs, Florida
  - Pfizer Investigational Site, Bradenton, Florida
  - Pfizer Investigational Site, Cape Coral, Florida
  - Pfizer Investigational Site, Fort Myers, Florida
  - Pfizer Investigational Site, Naples, Florida
  - Pfizer Investigational Site, Plantation, Florida
  - Pfizer Investigational Site, Port Charlotte, Florida
  - Pfizer Investigational Site, Sarasota, Florida
  - Pfizer Investigational Site, Venice, Florida
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Vincennes, Indiana
  - Pfizer Investigational Site, Ann Arbor, Michigan
  - Pfizer Investigational Site, Olive Branch, Mississippi
  - Pfizer Investigational Site, Oxford, Mississippi
  - Pfizer Investigational Site, Livingston, New Jersey
  - Pfizer Investigational Site, Asheville, North Carolina
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Collierville, Tennessee
  - Pfizer Investigational Site, Memphis, Tennessee
- Pfizer Investigational Site, Cologne, Germany

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=C016&StudyName=PF-3512676%20%28CPG%207909%29%20Injection%20For%20Patients%20Who%20Completed%20An%20Oncology%20Study%20Using%20PF-3512676%20%28CPG%207909%29